CLINICAL TRIAL: NCT03074630
Title: Dapagliflozin on Cholesterol Metabolism in DM2: Dissecting Its Effect on Dyslipidemia by Using Stable Isotope Based Cholesterol and Glucose Fluxes
Brief Title: Dapagliflozin and Cholesterol Metabolism in Type 2 Diabetes (DM2)
Acronym: DICE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, D van Raalte, PI, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: METC AMC 2016_016
Record Dates: First submitted 2016-06-22; First posted 2017-03-09 (Actual); Results first posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus, Type 2; Hypercholesterolemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypercholesterolemia | interventions — dapagliflozin; Rosuvastatin Calcium

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dapagliflozin 10mg and Rosuvastatin 10mg (Experimental): Rosuvastatin 10mg once daily for 9 weeks, with 5 weeks of once daily Dapagliflozin 10mg added
  Interventions: Drug: Dapagliflozin; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Dapagliflozin — 5 weeks 10mg dapagliflozin once daily
  Other Names: Forxiga
Drug: Rosuvastatin — 9 weeks 10mg dapagliflozin once daily
  Other Names: Crestor

SUMMARY:
Objective: To investigate the effect of 5 weeks dapagliflozin 10 mg once daily treatment on glucose and lipid fluxes in patients with type 2 diabetes.

Study design: Single center single arm (mechanistic) intervention trial.

Study Population: Male or postmenopausal female patients with type 2 diabetes BMI > 25 kg/m2and more than 12 weeks a stable dose of metformin treatment > 1500mg, HbA1C ≥6.5% - <8.5%, Fasting Plasma Glucose (FPG) <13.2 mmol/l, LDL cholesterol >2.5 mmol/l, willing to switch to rosuvastatin 10mg once daily for 4 weeks, and then receive 10 mg dapagliflozin once daily orally, for 5 weeks.

Treatment: After a statin washout fase of 4 weeks, baseline cholesterol synthesis will be measured (2H3 Leucine, 2H2O deuterated water). Then, treatment with rosuvastatin 10mg for 4 weeks will be initiated after which, patients will undergo glucose (2H2enriched glucose) and lipid flux (2H3 Leucine, 2H2O deuterated water and oral 1,2,3,4-13C16 - palmitate enrichment measurements) followed by 5 weeks treatment with dapagliflozin 10mg once daily. In the final week glucose/lipid flux measurements will be repeated.

Sample Size: 12 DM2 subjects.

Outcome measures: The primary endpoint is effect of 5 weeks Sodium-Glucose Linked co-transporter (SGLT) 2 inhibition on LDL cholesterol synthesis in patients with DM2. Secondary endpoints are effect of SGLT2 inhibition on triglyceride and cholesterol fluxes as well as (hepatic and peripheral) insulin sensitivity and energy expenditure. Finally, effect of SGLT2 inhibition on dietary intake, liver fat content (MRI liver) and fecal microbiome will be studied at these timepoints.

DETAILED DESCRIPTION:
Background: Type 2 diabetes is associated with an increased cardiovascular risk. Besides metformin, a new treatment strategy is oral SGLT2 inhibition (dapagliflozin), Although the recently published, first-in-class cardiovascular outcome trial (EMPA-REG OUTCOME) has suggested a beneficial effect on all cause cardiovascular mortality upon SGLT2 inhibition, a known (class) side effect in worsening of dyslipidemia in all DM2 patients. The investigators thus aim to dissect the effect of SGLT2 inhibition (Dapagliflozin 10mg once daily for 5 weeks) on glucose and lipid fluxes in uncomplicated DM2 subjects.

Objective: To investigate the effect of 5 weeks dapagliflozin 10 mg once daily treatment on glucose and lipid fluxes in patients with type 2 diabetes.

Study design: Single center single arm (mechanistic) intervention trial.

Study Population: Male or postmenopausal female patients with type 2 diabetes BMI > 25 kg/m2and more than 12 weeks a stable dose of metformin treatment > 1500mg, HbA1C ≥6.5% - <8.5%, FPG<13.2 mmol/l, LDL cholesterol >2.5 mmol/l, willing to switch to rosuvastatin 10mg once daily for 4 weeks, and then receive 10 mg dapagliflozin once daily orally, for 5 weeks.

Treatment: After a statin washout fase of 4 weeks, baseline cholesterol synthesis will be measured (2H3 Leucine, 2H2O deuterated water). Then, treatment with rosuvastatin 10mg for 4 weeks will be initiated after which, patients will undergo glucose (2H2enriched glucose) and lipid flux (2H3 Leucine, 2H2O deuterated water and oral 1,2,3,4-13C16 - palmitate enrichment measurements) followed by 5 weeks treatment with dapagliflozin 10mg once daily. In the final week glucose/lipid flux measurements will be repeated.

Outcome measures: The primary endpoint is effect of 5 weeks SLGT2 inhibition on LDL cholesterol synthesis in patients with DM2. Secondary endpoints are effect of SGLT2 inhibition on triglyceride and cholesterol fluxes as well as (hepatic and peripheral) insulin sensitivity and energy expenditure. Finally, effect of SGLT2 inhibition on dietary intake, liver fat content (MRI liver) and fecal microbiome will be studied at these timepoints.

Sample Size: Based on published data, the investigators expect 10% higher plasma LDL level (from 3.1 ± 0.8 to 1.7 ± 0.4 mmol/l ) upon SGLT2 inhibition in DM2. DM2 subjects have concomitant LDL- ApoB synthesis (1.8 ± 0.4 gram/day) after 4 weeks of rosuvastatin 10mg. Assuming an increase in LDL-apoB synthesis of 0.3 gram/day with SD of 0.4 and using single-sided test (with alfa of 0.05 and 85% power), the sample size needs to be 11 DM2 subjects on dapagliflozin 10mg treatment. Taking a 10% patient dropout rate, the aim is to include 12 DM2 subjects in total.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The risk for patients to participate in this study is minimal. All of the stable isotopes are GMP produced and analyses techniques have been previously used and published by the investigators. Also, REE and liver MRI measurements are not associated with adverse events. Both rosuvastatin and dapagliflozin have been approved by FDA/EMA and are widely prescribed. In total 470 ml blood (100 ml per lipidflux day, 90 ml per clamp day) will be drawn over period of 13 weeks (divided over 5 visits).

ELIGIBILITY:
Inclusion Criteria:

* Male or postmenopausal female patients ;
* Type 2 diabetes mellitus(HbA1C ≥6.5% - <8.5%)
* At least 12 weeks of stable dose metformin treatment, FPG<13.2 mmol/l
* LDL cholesterol >2.5 mmol/l
* Willing to switch used statin to rosuvastatin 10mg once daily
* 18-75 years of age
* Ability to provide informed consent

Exclusion Criteria:

* History of cardiovascular event
* Smoking
* exogenous insulin use
* Creatinin clearance < 60ml/min
* Alcohol abuse (>4 units/day)
* AST or ALT elevation (>2.5x upper limit)
* Contraindication to MR scanning (i.e. pacemaker, metallic foreign body, claustrophobia)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Max Nieuwdorp, MD/PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dapagliflozin: Dapagliflozin treatment for 5 weeks
Period: Overall Study
Arm/Group | Dapagliflozin
Started | 12
Completed | 11
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Dapagliflozin: Nine male and 3 postmenopausal female participants were included. One female participant was excluded during the study due to missing data, as we were unable to place a venous catheter during the second hyperinsulinemic clamp, thus we present the analysis for the 11 evaluable participtans.
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 64 [50 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma LDL Cholesterol
Description: Before and after 5 weeks of dapagliflozin on rosuvastatin background.
Time Frame: 5 weeks
Measure: Median (Full Range); unit: mmol/L
Groups:
- Dapagliflozin: 5 weeks of dapagliflozin
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 11
mmol/L | -0.1 [-0.2 to 0.2]

2. Secondary Outcome: Change in Plasma HDL Cholesterol
Description: Change in plasma HDL cholesterol following dapagliflozin
Time Frame: 12 weeks
Population: 5 weeks of dapagliflozin added to rosuvastatin
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 11
mmol/L | 0.08 [-0.03 to 0.13]

3. Secondary Outcome: Change in Total Cholesterol
Description: Change in total cholesterol following dapagliflozin
Time Frame: 5 weeks
Population: treated with 10mg dapagliflozin
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 11
mmol/L | -0.01 [-0.42 to 0.29]

4. Secondary Outcome: Change in Plasma Triglycerides
Description: Change in plasma Triglycerides following dapagliflozin
Time Frame: 5 weeks
Population: dapagliflozin treatment
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 11
mmol/L | 0.10 [-0.41 to 0.34]

5. Secondary Outcome: Change in Plasma FFA
Description: Change in plasma FFA following dapagliflozin
Time Frame: 5 weeks
Population: 5 weeks of dapagliflozin
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 11
mmol/L | 0.20 [0.04 to 0.78]

6. Secondary Outcome: Change in Cholesterol Fluxes
Description: Including cholesterol production, cholesterol excretion, cholesterol degradation. Before and after 5 weeks of dapagliflozin on rosuvastatin background.
Time Frame: 5 weeks
Population: These measurements were conditional, and have not been performed due to the absent change in the primary outcome.
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in Triglyceride Fluxes
Description: as for outcome 6
Time Frame: 5 weeks
Population: These measurements were conditional, and have not been performed due to the absent change in the primary outcome.
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 0

8. Secondary Outcome: Change in Peripheral Insulin Sensitivity
Description: Before and after 5 weeks of dapagliflozin on rosuvastatin background, measured as glucose disposal during hyperinsulinemic euglycemic clamp
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: umol/kg/min
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 11
umol/kg/min | 1.6 (10.7)

9. Secondary Outcome: Liver Fat MRI Spectrum
Description: Before and after 5 weeks of dapagliflozin on rosuvastatin background
Time Frame: 5 weeks
Population: This measurement was conditional, and has not been performed due to the absent change in the primary outcome. Liver fat content was not measured.
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 0

10. Secondary Outcome: Fecal Microbiome Composition
Description: Before and after 5 weeks of dapagliflozin on rosuvastatin background, different bacterial strains will be quantified in fresh fecal samples.
Time Frame: 5 weeks
Population: Sample collection failed. There were not enough samples to perform a proper analysis. Therefore, the few samples that were collected have not been measured and no data is available.
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 0

11. Secondary Outcome: Bile Salt Excretion
Description: Before and after 5 weeks of dapagliflozin on rosuvastatin background
Time Frame: 5 weeks
Population: This measurement was conditional, and has not been performed due to the absent change in the primary outcome. Since there was no change in plasma cholesterol, this was no longer interesting and samples were not measured
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 0

12. Secondary Outcome: Urinary Glucose Excretion
Description: Before and after 5 weeks of dapagliflozin on rosuvastatin background
Time Frame: 5 weeks
Population: Subtracted from glucose disposal rate, not separately analyzed in paper
Measure: Median (Full Range); unit: mg/min
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 11
mg/min | 44 [20 to 64]

13. Secondary Outcome: Urinary Sodium Excretion
Description: Before and after 5 weeks of dapagliflozin on rosuvastatin background
Time Frame: 5 weeks
Population: This measurement was conditional, and has not been performed due to the absent change in the primary outcome.
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 5 weeks
Description: Patient reported and actively assessed
Groups:
- Adverse Events: 5 weeks of dapagliflozin
Arm/Group | Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events (N=12)
genital fungal infection (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The comparatively small number of participants, the absence of a control group and short follow-up time limit the study and we only included subjects with uncomplicated type 2 diabetes on metformin monotherapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT03074630/Prot_SAP_000.pdf